CLINICAL TRIAL: NCT01039740
Title: Pharmacogenetic Study of Mirtazapine Response in Depressed Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Doh Kwan Kim, M.D., Ph.D., Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-08-092
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Depression
Keywords: Pharmacogenomics; Prediction of Mirtazapine response; Depressed patients; Mirtazapine response; Adverse event
MeSH Terms: conditions — Depression | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Responders (Experimental): Reponders is a patients group who showed 50% or greater decrease in the HAM-D score at 6 weeks after treating with mirtazapine
  Interventions: Drug: Mirtazapine
- Non-responders (Experimental): Non-responders is a patients group who did not show 50% or greater decrease in the HAM-D score at 6 weeks after treating with mirtazapine
  Interventions: Drug: Mirtazapine

INTERVENTIONS:
Drug: Mirtazapine — Mirtazapine administration for 6 weeks under therapeutic dose
  Other Names: Mirtazapine_Remeron, Avanza, Zispin

SUMMARY:
The purpose of this study is to determine whether pharmacogenetic study predict Mirtazapine responsiveness in advance before the appearance of the drug effect until 4-6 weeks after administration of Mirtazapine.

DETAILED DESCRIPTION:
The purpose of this study is

1. to determine whether genomic differences between drug responders and nonresponders predict the response of Mirtazapine and
2. to construct the prediction model for Mirtazapine treatment in depressed patients in order to aid to select the genetically matching drug.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible patients were enrolled in the clinical trials program of hte Samsung Medical Center Geropsychiatry and Affective Disorder Clinics(Seoul, Korea). They received a semistructured diagnostic interview, the Samsung Psychiatric Evaluation Schedule. The affective disorder section of the Samsung Psychiatric Evaluation Schedule uses the Korean version of the structured clinical interview for the diagnostic and statistical manual of mental disorders, Fourth edition.
2. interview with one more patient's family member for objective diagnosis and final diagnosis decision by agreements of two more psychiatric physicians

Exclusion Criteria:

1. received psychotropic medication within 2 weeks of the study or fluoxetine within 4 weeks
2. potential study participants for pregnancy, significant medical conditions, abnormal laboratory baseline values, unstable psychiatric features(eg.suicidal), history of alcohol of drug dependence, seizures, head trauma with loss of consciousness, neurological illness, or concomitant Axis I psychiatric disorder.

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2003-02; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Mirtazapine response at 2,4,6 weeks and adverse events (A/E) monitoring at 1,2,4,6 weeks | 6 weeks

SECONDARY OUTCOMES:
Biological value at 0 and 6 weeks | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Doh Kwan Kim, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Kangnam, Seoul, South Korea